CLINICAL TRIAL: NCT07183735
Title: A Crossover Trial to Examine the Efficacy of a Powder to Improve Sleep Quality and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beam (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20417
Record Dates: First submitted 2025-08-07; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Sleep; Sleep Disorder
Keywords: Sleep Quality
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEAM Dream Powder (Experimental)
  Interventions: Dietary Supplement: BEAM Dream Powder
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Control

INTERVENTIONS:
Dietary Supplement: BEAM Dream Powder — A powdered sleep supplement. Administered daily, mixed with 8-12 oz hot water, 30 minutes before bedtime during Weeks 3-6.
  Arms: BEAM Dream Powder
Dietary Supplement: Placebo Control — A powdered placebo product. Administered daily, mixed with 8-12 oz hot water, 30 minutes before bedtime during Weeks 1-2.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled crossover study to assess the efficacy of BEAM's Dream Powder in improving sleep health among 40 adults. Participants will use a placebo for 2 weeks, followed by the test product for 4 weeks, with sleep data collected via questionnaires and a Fitbit sleep tracker.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18+ years old
* Self-reported issues with sleeping, falling asleep, or staying asleep.
* Willing to discontinue any supplements, medications, herbal remedies, or melatonin products used to assist with sleep for the study duration.
* Willing to avoid introducing any other supplements, medications, herbal remedies, or melatonin products used to assist with sleep for the duration of this trial.
* Willing to maintain their standard sleep pattern and activity level for the duration of the study.
* Be generally healthy and not live with any uncontrolled chronic disease.

Exclusion Criteria:

* Diagnosed with any chronic sleep condition, including but not limited to insomnia, narcolepsy, or sleep apnea.
* Women who are pregnant, breastfeeding, or trying to conceive.
* Anyone unwilling or unable to follow the study protocol.
* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Is currently undergoing, or planning to undergo, any significant medical procedures during the study period.
* Has undergone any surgeries or invasive treatments in the last six months.
* A history of severe allergic reactions, including but not limited to any of the product's ingredients.
* Anyone with a nut allergy.
* Heavy drinkers. A heavy drinker is considered to be a woman who drinks 8 or more alcoholic drinks per week or a man who drinks 15 or more alcoholic drinks per week.
* Anyone who uses illicit drugs.
* Use any prescription medication, over-the-counter, or herbal remedies that can affect sleep.
* Have a job that involves working the third or night shifts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality as measured by the Sleep Quality Scale (SQS) | Baseline, Week 2, Week 4, Week 6
  Sleep quality will be assessed using the self-reported Sleep Quality Scale (SQS), a validated questionnaire evaluating subjective sleep quality.
Change in sleep quantity and architecture as measured by sleep tracker | Baseline, Week 2, Week 4, Week 6
  Objective sleep metrics (e.g., time to fall asleep, deep sleep, REM sleep, sleep transitions, sleep duration, and frequency of waking) will be collected using a sleep tracking device.

SECONDARY OUTCOMES:
Change in perceived restfulness as measured by self-reported questionnaire | Baseline, Week 2, Week 4, Week 6
  Participants will report perceived restfulness levels to assess subjective recovery and rest post-intervention.
Change in overall energy levels as measured by self-reported questionnaire | Baseline, Week 2, Week 4, Week 6
  Participants will rate their energy levels using a structured questionnaire.
Change in emotional well-being as measured by self-reported questionnaire | Baseline, Week 2, Week 4, Week 6
  Emotional well-being will be assessed using a validated self-report measure.
Change in cognitive function as measured by self-reported questionnaire | Baseline, Week 2, Week 4, Week 6
  Cognitive function will be assessed through a participant questionnaire evaluating attention, memory, and mental clarity.
Change in dietary behavior (e.g., hunger levels) as measured by self-reported questionnaire | Baseline, Week 2, Week 4, Week 6
  Participants will report perceived hunger levels and related dietary behavior using a structured questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States